CLINICAL TRIAL: NCT00465751
Title: Effects of Activation of the Farnesoid X Receptor (FXR) on Hepatic Lipid and Glucose Metabolism in Patients With the Metabolic Syndrome and Familial Forms of Hypertriglyceridemia
Brief Title: Effects of FXR Activation on Hepatic Lipid and Glucose Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKBB 211/04 SB
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Metabolic Syndrome; Familial Hypertriglyceridemia; Familial Combined Hyperlipidemia
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipoproteinemia Type IV; Hyperlipidemia, Familial Combined | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): chenodeoxycholic acid treatment
  Interventions: Drug: chenodeoxycholic acid
- B (Placebo Comparator): placebo treatment
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: chenodeoxycholic acid — chenodeoxycholic acid 500 mg capsules tid po
  Arms: A
Drug: placebo capsules — placebo capsules containing mannitol tid po
  Arms: B

SUMMARY:
The purpose of this study is to determine whether chenodeoxycholic acid decreases de novo hepatic lipogenesis, hepatic fat content, hepatic triglyceride production and plasma triglyceride concentrations and improves hepatic glucose metabolism in patients with the metabolic syndrome, Familial Hypertriglyceridemia and Familial Combined Hyperlipidemia.

DETAILED DESCRIPTION:
Insulin resistance has been found to be the key pathophysiological factor of the metabolic syndrome and may precede the onset of impaired glucose tolerance, diabetes and dyslipidemia. Recently, nonalcoholic fatty liver disease (NAFLD), has been identified as another feature of this syndrome. Importantly, a close relation between liver fat content and hepatic insulin sensitivity has been described. We hypothesize that activation of FXR with chenodeoxycholic acid decreases hepatic de novo lipogenesis and subsequently hepatic fat content and triglyceride production. The decrease in liver fat content will be associated with improved hepatic insulin sensitivity and a decrease in hepatic glucose production.

Patients diagnosed with metabolic syndrome, familial hypertriglyceridemia or familial combined hyperlipidemia will be recruited from the the outpatients department of the Division of Endocrinology, Diabetology and Clinical Nutrition, University Hospital Basel. Eligible patients will be admitted to the CRC for metabolic studies, including baseline blood samples for the measurement of hormones, cytokines and adipokines, euglycemic-hyperinsulinemic clamp studies for the assessment of glucose turnover and insulin sensitivity and in vivo NMR studies to determine intrahepatic and intramyocellular lipid content. Patients will alternatively receive chenodeoxycholic acid and placebo. The study population will be compared to a group of age, gender and weight matched normolipidemic controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. Patients with a metabolic syndrome defined by the presence of >= 3 of the following criteria:

   * Abdominal obesity (waist circumference > 102 cm in men, > 88 cm in women)
   * Fasting plasma triglycerides > 1.7 mmol/l
   * HDL cholesterol < 1.0 mmol/l in men and < 1.3 mmol/l in women
   * Blood pressure > 130/85 mmHg or antihypertensive medication
   * Fasting plasma glucose > 6.1 mmol/l
3. Patients with Familial Combined Hyperlipidemia characterized by the following criteria:

   * Fasting plasma triglycerides > 1.7 mmol/l
   * Fasting plasma apolipoprotein B concentrations > 1.2 g/l
   * Family history with hypertriglyceridemia and/or hypercholesterolemia present in at least 1 additional first degree family members
4. Patients with Familial Hypertriglyceridemia characterized by the following criteria:

   * Fasting plasma triglycerides > 2.3 mmol/l
   * Family history of hypertriglyceridemia in at least 1 additional first degree family member
   * Absence of the metabolic syndrome as defined above
5. Controls fulfilling the following criteria:

   * Non smoking.
   * No current or previous organ or systemic disease (including diabetes and lipid disorders).
   * Plasma triglycerides and cholesterol within the normal range (see exclusion criteria).
   * Plasma glucose concentrations <6.1 mmol/l Subjects meeting criterium 1 and any of the criteria 2. - 5. are eligible for the study.

Exclusion Criteria:

1. Any significant hepatic, cardiac, pulmonary, renal, neurological, musculoskeletal, hematological or endocrine disease.
2. Any form of primary or secondary hyperlipidemia other than the metabolic syndrome, FHTG or FCHL. [These may include: Familial hypercholesterolemia and Familial defective apolipoprotein B (to be assessed by family history and lipid profiles), and Familial Dysbetalipoproteinemia (to be assessed by apo E genotyping), hypothyroidism, nephrotic syndrome, diabetes mellitus, cholestatic liver disease, drug induced hyperlipidemia (thiazides > 25 mg/d, non cardioselective betablockers, isotretinoin, systemic glucocorticoids, cyclosporin A, tacrolimus, non nucleoside HIV protease inhibitors)].
3. Plasma TG levels > 12 mmol/l in the past or at any time point during the study.
4. History of acute pancreatitis
5. History of cardiovascular disease, i.e. coronary artery disease, cerebrovascular disease, peripheral vascular disease, when assessed by medical history, physical exam. Additionally, a stress test will be performed in subjects with MS and FCHL at risk for CHD (see below).
6. Pregnant or Breast Feeding women
7. Woman of childbearing potential not using a reliable method of birth control such as oral contraceptives or IUD.
8. Alcohol intake of greater than 1 drink daily.
9. Cigarette smokers
10. History of claustrophobia
11. Ferromagnetic implants including pacemakers.
12. Subjects refusing or unable to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10

PRIMARY OUTCOMES:
plasma triglyceride concentrations | 3 months

SECONDARY OUTCOMES:
hepatic insulin sensitivity | 3 months
heptic triglyceride content | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bilz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland